CLINICAL TRIAL: NCT05994001
Title: Two Stage, Multi-center Trial of Candonilimab in Combination With LM-302 for Treatment of Patients With Claudin 18.2 Positive-advanced Biliary Tract Cancer After Failure of Standard of Chemotherapy and PD1/PD-L1 Antibody
Brief Title: Candonilimab in Combination With LM-302 for Claudin 18.2 Positive-advanced Biliary Tract Cancer After Failure of Standard of Chemotherapy and PD1/PD-L1 Antibody
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSAB-Calm
Record Dates: First submitted 2023-07-21; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Biliary Tract Cancer; Candonilimab; Claudin 18.2
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Each cycle of the first phase was defined as cardonilizumab (6mg/kg,Q2W) combined with different concentrations of 1.6mg/kg or 1.8mg/kg LM-302 (Q2W), 14 days as a course of treatment, and the combined dose (RP2D) of LM-302 during combination therapy was determined according to the 3+3 design.
  In the second phase, Claudin18.2 expression was positive, and the positive population was randomly assigned to trial group 1, trial group 2, and trial group 3.
  Group 1:6 mg/kg cardonilizumab, 14 days for 1 course. Group 2:1.8mg /mg LM-302 was treated for 1 course for 14 days. Group 3: 6 mg/kg cardonilizumab for 14 days was a course of treatment; RP2D LM-302 is 1 course of treatment for 14 days.
Who Masked: Participant
Masking Description: Each cycle of the first phase was defined as cardonilizumab (6mg/kg,Q2W) combined with different concentrations of 1.6mg/kg or 1.8mg/kg LM-302 (Q2W), 14 days as a course of treatment, and the combined dose (RP2D) of LM-302 during combination therapy was determined according to the 3+3 design.
  In the second phase, Claudin18.2 expression was positive, and the positive population was randomly assigned to trial group 1, trial group 2, and trial group 3.
  Group 1:6 mg/kg cardonilizumab, 14 days for 1 course. Group 2:1.8mg /mg LM-302 was treated for 1 course for 14 days. Group 3: 6 mg/kg cardonilizumab for 14 days was a course of treatment; RP2D LM-302 is 1 course of treatment for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 6 mg/kg cardonilizumab, 14 days for 1 course.
  Interventions: Drug: cardonilizumab
- Group 2 (Experimental): 1.8mg /mg LM-302 was treated for 1 course for 14 days.
  Interventions: Drug: LM-302
- Group 3 (Experimental): 6 mg/kg cardonilizumab for 14 days was a course of treatment; RP2D LM-302 is 1 course of treatment for 14 days
  Interventions: Drug: cardonilizumab; Drug: LM-302

INTERVENTIONS:
Drug: cardonilizumab — cardonilizumab:PD1 and CTLA-4 bispecific antibody
  Other Names: PD1 and CTLA-4 bispecific antibody
  Arms: Group 1; Group 3
Drug: LM-302 — LM-302 :ClAUDIN 18.2-ADC
  Other Names: ClAUDIN 18.2-ADC
  Arms: Group 2; Group 3

SUMMARY:
In this clinical study, we will evaluate the efficacy and safety of cardonilimumab (PD1 monoclonal antibody and CTLA-4 monoclonal antibody bisspecific antibodies) and LM-302 (Claudin18.2-ADC) in Claudin18.2-positive advanced BTC patients who have progressed after SOC and PD1/PD-L1 monoclonal antibody treatment.

DETAILED DESCRIPTION:
The prognosis for unresectable and metastatic biliary malignancies (BTC) is extremely poor, with a median overall survival of only about 1 year for advanced biliary tumors treated with gemcitabine and cisplatin or combined with duvaliumab (PD-L1) as recommended by NCCN guidelines. At present, the NCCN guidelines recommend that the posterior line treatment of advanced BTC, such as FOLFOX, has a very limited effect, with an objective response rate of only about 5% and a median survival time of only about 6 months. There is an urgent need to develop new therapeutic methods to improve patient survival. Chronic inflammation caused by viral infection and bile duct stones are the most common potential risk factors for BTC, and immune system abnormalities play a key role in the occurrence and development of BTC. BTC, including intrahepatic cholangiocarcinoma (iCCA), showed abnormal expression of immune checkpoint molecules PD-L1 and CTLA-4 and obvious heterogeneity. Therefore, immunotherapy is of great value. TOPAZ-1 and KENOTE-966 studies both showed the value of PD-L1/PD1 monoclonal antibody in the treatment of advanced BTC. There is currently a lack of treatment options for progression after treatment with standard chemotherapy (SOC) combined with PD-L1/PD1 monoclonal antibodies. CTLA-4 inhibitors combined with PD-1/PD-L1 inhibitors have shown significantly enhanced clinical effects. Clinical studies on treating CTLA-4 inhibitors combined with PD-1/PD-L1 inhibitors have been carried out in several solid tumors. Although significant therapeutic effects have been achieved, adverse reactions (AEs) that cannot be ignored limit the benefit of patients. Claudin18.2 is a newly discovered tumor therapeutic target. Multiple clinical studies have shown that Claudin18.2 monoclonal antibody, Claudin18.2-ADC, and Cart-Claudin18.2 have good ORR in Claudin18.2-positive gastric cancer. At present, no independent research data on advanced BTC has been reported.

In this clinical study, we will evaluate the efficacy and safety of cardonilimumab (PD1 monoclonal antibody and CTLA-4 monoclonal antibody bispecific antibodies) and LM-302 (Claudin18.2-ADC) in Claudin18.2-positive advanced BTC patients who have progressed after SOC and PD1/PD-L1 monoclonal antibody treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced BTC that is not resectable or metastatic or recurred after surgery, histologically confirmed, and sufficient tissue specimens are provided for PD-L1, CTLA-4, Claudin18.2 immunohistochemistry and exon sequencing. Claudin18.2 expression is not required at the first stage. In the second stage, Claudin18.2-positive patients were required to be enrolled (≥40% immunohistochemical expression of Claudin18.2 was considered positive, <40% was considered negative, and two independent pathologists made the judgment. If there was any discrepancy, the third pathologist was asked to make the judgment together).
2. Failure of standard chemotherapy (gemcitabine or platinum or fluorouracil) and PD1/PD-L1 for advanced BTC due to disease progression or toxicity;
3. Measurable lesions;
4. For patients with a prior history of hepatic chemoembolization, radiofrequency ablation/intervention, or radiotherapy, measurable lesions outside the chemoembolization or radiotherapy area or measurable progression lesions at the chemoembolization or radiotherapy site must be present;
5. ECOG physical state ≤ 2;
6. Life expectancy > 3 months;
7. Adequate renal function: creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or glomerular filtration rate (GFR) ≥ 60mL/min/ 1.73m2;
8. Adequate liver function: bilirubin ≤ 1.5 × ULN and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN;
9. Adequate bone marrow reserve: absolute value of neutrophil (ANC) > 1500/mcl, platelets (Plts) > 75,000/mcl, hemoglobin (Hgb) ≥ 9.0g/dl;
10. Prothrombin time/activated partial thromboplastin time (PT/PTT) <1.5 × ULN;
11. Age ≥18 years old, male or female;
12. Participants with a prior history or persistent hepatitis C virus (HCV) infection will be eligible to participate in the study. Participants receiving antiviral therapy must complete treatment at least 1 month before the start of the study intervention. For HCV subjects who have not received or have not completed antiviral therapy, treatment should be initiated only after liver function has remained stable for at least 3 months during the study intervention.
13. Hepatitis B controlled subjects are eligible to participate in the study as long as they meet the following criteria:

    Subjects with chronic hepatitis B virus (HBV) infection (defined as hepatitis B surface antigen [HBsAg] positive and/or detectable HBV DNA) must have a HBV viral load of less than 2000 IU/ml prior to first dosing of the study intervention or a 10-fold reduction in HBV viral load with antiviral therapy. Subjects treated with active HBV with a viral load below 2000 IU/ml should receive antiviral therapy throughout the study intervention.
14. Subjects who are clinically cured of HBV infection (defined as HBsAg negative and anti-HBC positive) and whose HBV viral load is not detectable at screening should have their HBV viral load checked every 8 weeks and should be treated for HBV if the viral load exceeds 2000 IU/ml. Antiviral therapy after completion of the study intervention should follow local guidelines.

Exclusion Criteria:

* 1) Previous treatment with checkpoint inhibitor CTLA-4 monoclonal antibody, targeting Claudin18.2; 2) Major surgery or radiotherapy or intervention or ablation within 4 weeks before enrollment; 3) Active, known, or suspected autoimmune disease; 4) Congestive heart failure or symptomatic coronary artery disease within 3 months prior to enrollment; 5) Cerebrovascular accident occurred within the past 6 months; 6) Clinically significant bleeding, bleeding event, or thromboembolic disease within 6 months; 7) History of intestinal perforation; 8) Have a history of (non-infectious) pneumonia requiring steroid treatment or currently have pneumonia; 9) Known history of human immunodeficiency virus (HIV) infection; 10) A history of severely impaired lung function or interstitial lung disease; 11) Concurrent malignancies (other than adequately treated non-melanoma skin cancer, superficial transitional cell carcinoma of the bladder and cervical carcinoma in situ [CIS]) or any currently active malignancies have been diagnosed within the last 5 years; 12) Past or current evidence indicates any condition, treatment, or laboratory abnormality that may confuse the study results, interfere with the subject's participation throughout the study, or the investigator determines that participation in the study is not in the subject's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR(Phase II) | 24months
  Objective response rate (ORR) in patients with Claudin18.2-positive treated with cardonillizumab combined with LM302 (RECIST 1.1)(Phase II)
Incidence of Treatment-Emergent Adverse Events(Phase I) | 24months
  Safety of cardonilizumab in combination with different doses of LM-302 in patients with advanced BTC

SECONDARY OUTCOMES:
DOR | 24months
  duration of overall response
DCR | 24months
  disease control rate
OS | 24months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Oh DY, Lee KH, Lee DW, Yoon J, Kim TY, Bang JH, Nam AR, Oh KS, Kim JM, Lee Y, Guthrie V, McCoon P, Li W, Wu S, Zhang Q, Rebelatto MC, Kim JW. Gemcitabine and cisplatin plus durvalumab with or without tremelimumab in chemotherapy-naive patients with advanced biliary tract cancer: an open-label, single-centre, phase 2 study. Lancet Gastroenterol Hepatol. 2022 Jun;7(6):522-532. doi: 10.1016/S2468-1253(22)00043-7. Epub 2022 Mar 9. PMID 35278356